CLINICAL TRIAL: NCT02610374
Title: Diet / Gut Microbiome Interaction and Influence on Inflammatory Disease in HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-1692
Record Dates: First submitted 2015-10-23; First posted 2015-11-20 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: HIV
Keywords: Gut microbiota composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Other): HIV-positive individuals will be randomized to receive either an Agrarian diet or a Western-type diet for 4 weeks.
  Interventions: Other: Agrarian Diet; Other: Western-type Diet
- Cohort B (Other): HIV-negative high-risk individuals will be randomized to receive either an Agrarian diet or a Western-type diet for 4 weeks.
  Interventions: Other: Agrarian Diet; Other: Western-type Diet
- Cohort C (Other): HIV-negative low-risk individuals will be randomized to receive either an Agrarian diet or a Western-type diet for 4 weeks.
  Interventions: Other: Agrarian Diet; Other: Western-type Diet

INTERVENTIONS:
Other: Agrarian Diet — A diet higher in carbohydrates and lower in fats and sugars
Other: Western-type Diet — A diet higher in fats and lower in carbohydrates

SUMMARY:
The primary objective is to assess the effect of short-term diet modification on the microbiome composition, and inflammatory/metabolic disease markers in Antiretroviral therapy (ART)-treated HIV-infected participants and Human immunodeficiency virus (HIV)-negative controls in the United States.

DETAILED DESCRIPTION:
This is a randomized clinical trial. Fifty (50) Antiretroviral therapy (ART)-treated Human immunodeficiency virus (HIV) positive participants, 24 HIV negative controls matched for age and sex, and 24 HIV negative controls from a population at high risk for contracting HIV will be recruited into 3 cohorts. All participants will undergo a 4 week diet modification and will be randomly assigned to receive either an Agrarian diet or a Western-type diet. For the first 2 weeks, food will be provided to the participant, followed by an additional 2 weeks where participants will be provided a diet menu with recipes to prepare themselves. There will be 4 study visits and participation will last for up to 2 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected cohort (Cohort A)

  * Documentation of HIV-1 infection defined as a positive antibody test or plasma HIV-1 RNA (ribosomal ribonucleic acid).
  * Treated with ART (minimum of three antiretroviral drugs in regimen) for at least 12 months with no changes in antiretroviral drugs over the past 6 months
  * Plasma HIV-1 RNA ≤ 50 copies/mL in the preceding 6 months.
* HIV-negative cohorts (Cohort B and C)

  * Documentation of a negative HIV-1 antibody test
* All Cohorts

  * Age 18 to 65 years
  * Body mass index between 21-29 kg/m2 (non-obese)
  * Stable weight for at least 3 months (≤15% change in body weight)
  * Negative pregnancy test (if female)

Exclusion Criteria:

* Use of systemic (oral or parenteral) antibiotics within two months prior to study entry
* Active chronic infection such as hepatitis B or C or an active malignancy that requires systemic chemotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Change in plasma IL-6 concentration (All Participants) | 4 weeks
  - The change in plasma IL-6 from baseline to week 4 for all participants (Cohorts A, B & C) assigned to the Agrarian diet group will be compared to participants assigned to the Western diet group.
Change in plasma IL-6 concentration (HIV-Infected Participants) | 4 weeks
  - The change in plasma IL-6 from baseline to week 4 for HIV-infected participants (Cohort A) assigned to an Agrarian diet will be compared to HIV-uninfected participants (Cohort B & C) assigned to an Agrarian diet.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lozupone, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] O'Connor JB, Fouquier J, Neff CP, Sterrett JD, Marden T, Fiorillo S, Siebert JC, Schneider J, Nusbacher N, Noe AT, Fennimore B, Higgins J, Campbell TB, Palmer BE, Lozupone C. Agrarian diet improves metabolic health in HIV-positive men with Prevotella-rich microbiomes: results from a randomized trial. mSystems. 2025 Dec 17;10(12):e0118525. doi: 10.1128/msystems.01185-25. Epub 2025 Nov 26. PMID 41294355